CLINICAL TRIAL: NCT03732989
Title: Experimental Study Testing the Self-regulation Effects of a Social Assistive Robot Prototype During Moments of Emotional Stress
Brief Title: Testing Self-regulation Effects of a 'Smart Toy'
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Anna Freud National Centre for Children and Families (Other); University of California Santa Cruz (Other); Committee for Children (USA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3923/005
Record Dates: First submitted 2018-10-02; First posted 2018-11-07 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be aware of the other condition, i.e., that the device could be interactive/non-interactive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Non-interactive toy prototype (Active Comparator): 30 children will be given the same toy as participants in the experimental group, but without the interactive features (haptic feedback).
  Interventions: Device: Non-interactive toy prototype
- Experimental: Interactive toy prototype (Experimental): 30 children will be given the same toy as participants in the control group, but with the interactive features (haptic feedback).
  Interventions: Device: Interactive toy prototype

INTERVENTIONS:
Device: Interactive toy prototype — The interactive toy prototype takes the form of a hand-crafted plush toy, which was designed to support in-the-moment calming down strategies. The interaction relies on a number of sensors embedded in the 'creature' that register haptic interactions with the toy. In addition, a small vibration motor is used to indicate the creature's state by mimicking a frantic 'heartbeat'. If the creature is calming down in response to the child's touching of the sensors, the heartbeat slows down and eventually turns into happy purring (cf. paper linked below for more details about the design process).
  Arms: Experimental: Interactive toy prototype
Device: Non-interactive toy prototype — This toy is the same as the interactive one, but with the interactivity features (haptic feedback) turned off so that it looks and feels like a regular, hand-crafted plush toy.
  Arms: Control group: Non-interactive toy prototype

SUMMARY:
The present experimental study aims to explore the effect of an interactive smart toy on children's stress modulation during a stressful experience compared to a non-interactive prototype. It is expected that children given the interactive prototype will experience faster and more effective stress modulation, in comparison to those being given the non-interactive prototype.

These findings will complement the ecologically valid data from week-long at-home deployments of the interactive prototype with families with low socioeconomic status.

DETAILED DESCRIPTION:
The proposed experimental design relies on an established task that can induce a short-term stress response to enable us to the test of efficacy of the smart toy in helping children regulate their emotions in controlled settings. The investigators will use an adapted version of the well-established Trier Social Stress Test for Children (TSST-C). The TSST-C was chosen as it is one of the most popular and standardised methods to induce a strong psychosocial stress response in experimental settings, due to its socio-evaluative character and uncontrollability. Prior literature shows that (i) the TSST-C is suitable for children in our age range; and (ii) stress returns to normal levels shortly after children receive positive feedback from the experimenters.

The original TSST-C protocol consists of a preparation period, public speaking task and mental arithmetic task. The investigators have chosen to only use the preparation period, public speaking task and anticipation of the mental arithmetic task as stressors, as pilots suggest that these suffice to elicit a strong-enough stress response that will allow us to test the toy's efficacy; and it would be unethical to subject children to unnecessary tasks.

== Study protocol: ==

On arrival to the room where the experiment will take place, children in both groups will be informed that there are three tasks involved in the study:

1. giving a speech,
2. a calculation task, and
3. helping a newly discovered creature (the toy) which appears to be anxious calm down.

The children will then be fitted with the Empatica E4 wristband which will continuously and non-intrusively monitor their heart rate and skin conductance, and introduced to the toy in order to limit the impact of the novelty effect associated with it. Participants in the control group will be asked to imagine that the toy is a creature which is anxious, while participants in the experimental group will also be told that the creature's heartbeat is fast when it is anxious and slows down when it calms down. The researcher will demonstrate three soothing interactions with the toy (cuddling, stroking, and slow breathing) for 30 seconds and then give the children the toy for 1 minute, after which it will be returned to the researcher.

Following this introduction, participants will stay in the room for 10 minutes reading pictures books if they would like to in order to establish baseline stress levels. After 10 minutes have passed, the researcher will administer the state anxiety scale of the State Trait Anxiety Inventory for Children (STAI-CH).

Participants will then hear the beginning of a story and will be asked to finish it in a manner as exciting as possible in front of a microphone and a camera. Participants will be told that other study participants will do the same and will be prompted to perform better than them, even though in reality they will not be judged for their performance. Participants will remain in the room for 5 minutes preparing their story.

After the preparation period the researcher will administer the state anxiety scale for the second time. Following this, participants will be asked to stand in front of the microphone, the camera and the researcher, and finish the story as excitingly as possible in 3 minutes. If the participant finishes the story in less than 3 minutes, the researcher will ask them to continue in a friendly, supportive manner for a maximum of 3 times, using lines like "You are doing very well. You have to continue for a little bit longer, there is still more time to say your story."

After the speech task is completed the researcher will administer the state anxiety scale for the third time. Following this, the researcher will tell participants that it is time for the calculation task, which will supposedly be asking them to mentally subtract by 7's from a three-digit number. After saying this, the researcher will pretend that there are some issues with the camera that need to be fixed before they can start, and that they will have to shift the order of the two remaining tasks so that they have more time to fix the camera. At this point children will be exposed to one of the two conditions (interactive or non-interactive toy) for 5 minutes, following which they will complete the state anxiety scale for the final time.

The researcher will then tell children that due to the technical issues and time constraints they will not have to do the calculation task, but can rather move on to the last part of the study which is a 10-minute debriefing and feedback session. Every child will be told that they performed extremely well and that the experimenters pretended that they competing with the other participants to induce competitive conditions. The debriefing session will include a manipulation check (how stressfully the experienced the preparation period, speech task and anticipation of mental arithmetic task period) and a short interview about their experience, which will be audio-recorded.

At the end of the procedure, children will be allowed to relax in the room for 15 minutes. The researcher will suggest that they play with the interactive toy; sit down and take deep breaths; listen to guided mindfulness sessions; or read one of the age-appropriate books in the room.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7-10 years
* Understand English sufficiently to take part and complete study materials

Exclusion Criteria:

* Aged <7 years or >10 years
* Does not understand English sufficiently to take part and complete study materials

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of change in scores on the State Anxiety subscale of the State-Trait Anxiety Inventory for Children (STAI-CH; Spielberger, 1973) between the groups | 4 timepoints during a single study visit: (i) baseline ; (ii) right before participants are asked to perform the speech task; (iii) right after the speech task; and (iv) right after the 5-minute exposure to one of the two conditions
  The STAI-CH is a widely used instrument for measuring anxiety in children. The state subscale consists of 20 items which measure anxiety as a fleeting emotional state. Each STAI-CH item is a 3-point rating scale for which values of 1, 2, or 3 are assigned for each of the three alternative choices. Thus, scores on the subscale can range from a minimum of 20 to a maximum score of 60. Higher scores indicate greater anxiety.
Comparison of change in physiological stress levels between the groups | Continuously from baseline until the end of the experimental session (approximately 1 hour).
  Physiological stress reactivity will be measured by an Empatica E4 wristband which will continuously and non-intrusively monitor participants' heart rate and electrodermal activity throughout the experimental session. The change in physiological stress levels between the preparation for the speech task and post-exposure to one of the two conditions will be compared between the two participant groups.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Slovak, PhD, Principal Investigator — University College London; Anna Freud National Centre for Children and Families
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No